CLINICAL TRIAL: NCT02738580
Title: Analysis of Follicular Steroid Synthesis During Controlled Ovarian Stimulation With Recombinant FSH vs HMG in GnRH Antagonist Cycles
Brief Title: Follicular Steroid Genesis in Controlled Ovarian Stimulation
Acronym: ESTEFOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1512-VLC-066-EB
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Infertility; Controlled Ovarian Hyperstimulation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rFSH (Active Comparator): Controlled ovarian hyperstimulation with GnRH antagonists and rFSH in women with normal ovarian function.
  Interventions: Drug: COS with GnRH antagonists and rFSH
- HP-HMG (Active Comparator): Controlled ovarian hyperstimulation with GnRH antagonists and HP-HMG with normal ovarian function.
  Interventions: Drug: COS with GnRH antagonists and HP-HMG

INTERVENTIONS:
Drug: COS with GnRH antagonists and rFSH — Controlled ovarian hyperstimulation with GnRH antagonists and rFSH in women with normal ovarian function.
  Other Names: GnRH antagonists and rFSH
  Arms: rFSH
Drug: COS with GnRH antagonists and HP-HMG — Controlled ovarian hyperstimulation with GnRH antagonists and HP-HMG in women with normal ovarian function.
  Other Names: GnRH antagonists and HP-HMG
  Arms: HP-HMG

SUMMARY:
Serum concentrations of the different hormones involved in follicular steroid genesis during a cycle of controlled ovarian stimulation with recombinant FSH or HMG will be compared in this study. Serum Progesterone (P) levels at the end of Controlled Ovarian Stimulation (i.e. the day of triggering) have been related to cycle outcome, in terms of ongoing pregnancy and live birth rates. Large cohort studies show that P levels above a certain threshold are associated with poorer cycle outcome. The mechanisms behind P elevation are not well understood yet. It has been shown that P levels are positively related to ovarian response and to the dose of FSH given during COS. Furthermore, it has been well documented that P levels at the end of stimulation are significantly higher when recombinant (r) FSH is used for COS when compared to HMG, either in a GnRH agonist long protocol or in a GnRH antagonist protocol. Some authors suggest that this finding is explained by the fact that COS with rFSH provides a higher oocyte yield than when hMG is given, so the higher P levels observed would be explained by the larger number of follicles developed when rFSH is used. On the other hand, other authors explain this event by a different follicular esteroidogenesis when HMG is used for COS compared to rFSH The hypotheisis behind this assumption is that rFSH enhances P synthesis from its precursor pregnenolone in the granulosa cells. This P is unable to be further metabolized into androgens because of the lack of 17-20 lyase in the human granulosa cells, and therefore is delivered into circulation. On the other hand, when HMG is given for COS, the ∆4 pathway is promoted, and pregnenolone will be catabolized in to Dehidroepiandrostenodione (DHEA), in the theca cells, and this one to Androstenodione, which will be finally aromatized in to estrogens. This mechanism will explain the lower P and higher E2 levels observed in HMG cycles in comparison to rFSH cycles.

ELIGIBILITY:
Inclusion Criteria:

* Good physical and psychological condition
* Normal menstrual cycle (25-35 days)
* Normal ovarian reserve defined by serum ANH010-30 pMol/L
* All other criteria to fulfill by oocyte donors

Exclusion Criteria:

* Kidney failure
* Ovarian Polyquistic syndrome
* Any systemic or metabolic disfunction that counter indicates the use of gonadotrophins
* Any other reason that involves exclusion of the oocyte donation program

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Bosch, MDPhD, Principal Investigator — IVI VALENCIA
Locations (1):
- IVI Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosch E, Alama P, Romero JL, Mari M, Labarta E, Pellicer A. Serum progesterone is lower in ovarian stimulation with highly purified HMG compared to recombinant FSH owing to a different regulation of follicular steroidogenesis: a randomized controlled trial. Hum Reprod. 2024 Feb 1;39(2):393-402. doi: 10.1093/humrep/dead251. PMID 38037188

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rFSH | HP-HMG
Started | 56 (56 patients were assigned to this arms.) | 56
Completed | 52 (3 cycles cancelled due to por response to stimullation. 1 cycle cancelled due to SAE.) | 52 (2 cycles cancelled due to por response to stimullation 1 patient withdrawal 1 excluded)
Not Completed | 4 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — EXCLUDED FROM DONNOR PROGRAM | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rFSH | HP-HMG | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 56 | 112
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: SERUM PROGSTERONE CONCENTRATION
Description: Compare hormonal blood serum concentrations of progesterone during ovarian stimulation implied in follicular steroidogenesis during a cycle of Controlled Ovarian Stimulation with either r-FSH or HP-HMG.
Time Frame: 21 days
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | rFSH | HP-HMG
Number analyzed (Participants) | 52 | 52
ng/mL | 0.74 [0.22 to 1.26] | 0.45 [0.19 to 0.71]
Statistical Analysis 1: Comparison: rFSH vs HP-HMG; Test type: Superiority; p < 0.05, t-test, 2 sided — The proportion of patients with elevated Progesterone on last day of stimulation(>1.5 ng/mL) was compared between both groups using the Chi-square test; Mean Difference (Final Values) = 0.29, Standard Deviation 0.26

2. Primary Outcome: OVARIAN RESPONSE
Description: NUMBER OF FOLICLES REACHED AND PUNCTURED AFTER CONTROLED OVARIAN STIMULATION
Time Frame: 21 days
Measure: Mean (95% Confidence Interval); unit: folicles
Arm/Group | rFSH | HP-HMG
Number analyzed (Participants) | 52 | 52
folicles | 16.5 [9 to 24] | 17.5 [9.6 to 25.4]
Statistical Analysis 1: Comparison: rFSH vs HP-HMG; Test type: Superiority; p < 0.49, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 21 Days
Description: Coagulation panel alteration.
Arm/Group | rFSH | HP-HMG
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFSH (N=56) | HP-HMG (N=56)
COAGULATION PANEL ALTERATION (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — PT: 15,4 seg; INR: 1,3; Quick Index: 69%; TTPA: 38 seg. Hemmatic parameters at minimum normal limits She was reffered to hemathologist department. There was not more information about patient since january 2018.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT02738580/Prot_SAP_000.pdf